CLINICAL TRIAL: NCT05446831
Title: Efficacy and Safety of Baricitinib for Steroid-resistant/Relapse Immune Thrombocytopenia: A Single-arm, Open-label Phase II Study
Brief Title: Baricitinib for Steroid-resistant/Relapse Immune Thrombocytopenia
Acronym: BAITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-ITP2207
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: ITP; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Oral baricitinib was given at a dose of 4 mg daily for 6 months. Treatment was discontinued if very severe or life-threatening adverse events developed or at the patients' request.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Oral baricitinib was given at a dose of 4 mg daily. The decision to initiate rescue therapy was made after assessment of the extent of bleeding, patient preferences, lifestyle and activity, the complications of specific therapies, comorbidities that predisposed patients to bleeding and the tolerance of side effects. If a platelet count over 300,000/μL was observed for two consecutive tests at least 2 weeks apart, baricitinib treatment was interrupted.

SUMMARY:
Single-arm, open-label, single-center study to evaluate the efficacy and safety of baricitinib for the treatment of adults with steroid-resistant/relapse immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a prospective trial of 20 adults with ITP in China. Baricitinib is administered as 4 mg po. daily. Safety outcomes and efficacy outcomes are assessed on scheduled study visits (primary endpoint defined as durable response at 6-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia
2. Patients with chronic low platelet count (<30,000/μL) for 6 months who have failed at least one treatment for chronic low platelet count
3. Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation
4. Patients with a platelet count <30,000/μL or a platelet count <50,000/μL with clinically significant bleeding symptoms at the enrollment
5. Over 18 years old
6. Willing and able to provide written informed consent, and agreeable to the schedule of assessment

Exclusion Criteria:

1. Secondary immune thrombocytopenia (e.g. patients with HIV, HCV, Helicobacter pylori infection or patients with confirmed autoimmune disease)
2. Active or a history of malignancy
3. Pregnancy or lactation
4. Current or recent (<4 weeks prior to screening) clinically serious viral, bacterial, fungal, or parasitic infection
5. A history of symptomatic herpes zoster infection within 12 weeks prior to screening
6. Active or chronic viral infection from hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
7. Have evidence of active tuberculosis (TB), or have previously had evidence of active TB and did not receive appropriate and documented treatment, or have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB
8. Have experienced a clinically significant thrombotic event within 24 weeks of screening or are on anticoagulants and in the opinion of the investigator are not well controlled
9. Myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure
10. A history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data
11. Any of the following specific abnormalities on screening laboratory tests:

1) ALT or AST >2 x ULN, or total bilirubin ≥1.5 x ULN 2) hemoglobin <9 g/dL, or total white blood cell (WBC) count <2,500/µL, or neutropenia (absolute neutrophil count <1,200/µL), or lymphopenia (lymphocyte count <750/µL) 3) eGFR <50 mL/min/1.73 m^2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Durable response | 6 months
  The maintenance of a platelet count ≥30,000/μL, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
Complete response (CR) | 1 month
  Complete response (CR) was defined as a platelet count over 100,000/μL and absence of bleeding.
Response (R) | 1 month
  Response (R) as a platelet count over 30,000/μL and at least 2-fold increase of the baseline count and absence of bleeding.
Time to response | 6 months
  The time from starting treatment to time of achievement of CR or R.
Duration of response | 6 months
  Duration of response at 6-month follow up.
Early response | 7 days
  Achievement of CR or R at day 7
Initial response | 28 days
  Achievement of CR or R at day 28
Bleeding events | From the start of study treatment (Day 1) to the end of week 24
  Clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale.
Health-related quality of life (HRQoL) | From the start of study treatment (Day 1) to the end of week 24
  ITP-PAQ is used to assess the Health Related Quality of Life (HRQoL) before and after treatment.
Adverse events | From the start of study treatment (Day 1) to the end of week 24
  Adverse events (AEs) are reported and graded in accordance with the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China